CLINICAL TRIAL: NCT04220606
Title: Glutamate Concentrations in the Brain Over the Course of a Migraine-like Attack
Brief Title: 1H Magnetic Resonance Spectroscopy in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government); European Commission (Other)
Responsible Party: Principal Investigator, G.M. Terwindt, MD, Associate professor, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P07079.6
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Migraine Disorders; Migraine Without Aura; Headache Disorders, Primary; Headache Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Headache Disorders, Primary; Headache Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine without aura subjects (Other): Drug: Glyceryl trinitrate (GTN)
  Interventions: Drug: Glyceryl trinitrate (I.V. infusion 0.5 µg/kg/min over 20 min)
- Healthy subjects (Other): Drug: Glyceryl trinitrate (GTN)
  Interventions: Drug: Glyceryl trinitrate (I.V. infusion 0.5 µg/kg/min over 20 min)

INTERVENTIONS:
Drug: Glyceryl trinitrate (I.V. infusion 0.5 µg/kg/min over 20 min)

SUMMARY:
To investigate the glutaminergic system in the onset of migraine-like attacks.

DETAILED DESCRIPTION:
Glyceryl trinitrate infusion (GTN) is used to provoke migraine-like attacks in female migraine without aura patients. Apart from migraine without aura patients healthy female controls are also included as a control group. Over the course of a single day these females (migraineurs and healthy controls) were scanned three times on fixed time slots: before GTN infusion (baseline), 90 minutes and 270 minutes after start of GTN infusion. Scans are acquired on a 7 tesla scanner (Philips, Cleveland, USA) on software release 3 using a 32 channel receive array using single-volume proton magnetic resonance spectroscopy (1H MRS) with a volume of interest in the visual cortex glutamate, in which glutamate, GABA and other metabolites will be assessed. The primary endpoint; glutamate level changes towards the pre-ictal and ictal state with other metabolite (e.g. glutamine and GABA) changes as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine without aura according to the International Classification of Headache Disorders (ICHD)-3 beta criteria from 2013.
* At least one migraine attack per month in the preceding six months

Exclusion Criteria:

* Other neurological disorders apart from migraine
* Chronic medication apart from oral contraceptives
* Migraine with aura
* Chronic migraine with 15 or more headache days per month/with 8 or more migraine days per month
* Medication-overuse headache (ICHD-3 beta criteria)
* Women who are breastfeeding, pregnant, or planning to become pregnant
* Contra-indications for 7 tesla MRI scanner
* Contra-indications for GTN administration (e.g. nitrate allergy, heart condition)
* Healthy controls (with no first degree relative with migraine or trigeminal autonomic cephalalgia)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Glutamate | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in glutamate level

SECONDARY OUTCOMES:
Glutamine | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in glutamine level
GABA | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in GABA level
N-acetylaspartate | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in N-acetylaspartate level
Phosphoethanolamine | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in phosphoethanolamine level
Myo-inositol | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in myo-inositol level
Glutathione | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in glutathione level
Aspartate | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in aspartate level
Creatine | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in creatine level
Choline | From baseline towards the pre-ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) and ictal (assessed at 90 and/or 270 minutes after GTN depending on clinical condition) state
  Changes in choline level

IPD SHARING:
Plan to Share IPD: No